CLINICAL TRIAL: NCT01537614
Title: Pharmacokinetic Study of Aerosolized Colimycin in Cystic Fibrosis
Acronym: COLI-VLM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COLI-VLM
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

ARMS (2):
- COLIMYCINE injectable (Experimental)
  Interventions: Drug: COLIMYCINE injectable
- COLIMYCINE inhalation (Experimental)
  Interventions: Drug: COLIMYCINE inhalation

INTERVENTIONS:
Drug: COLIMYCINE inhalation — 2 MILLION UI
  Arms: COLIMYCINE inhalation
Drug: COLIMYCINE injectable — 2 MILLIONS UI
  Arms: COLIMYCINE injectable

SUMMARY:
Pharmacokinetics of colimycin will be assessed during 12 hours after administration of 2M UI colimycin either as an aerosol or after IV injection, the administration being separated by 5 to 10 days intervals

ELIGIBILITY:
Inclusion Criteria:

* Males and females, adults.
* Suffering from stable cystic fibrosis
* Colonized by P. aeruginosa
* Having given informed consent.
* Able to follow the protocol
* Having a social insurance

Exclusion Criteria:

* Renal insufficiency
* Allergy to colistin or polymixins
* Myasthenia
* Recent severe hemoptysis
* Liver cirrhosis and hepatic insufficiency
* Hypoalbuminemia
* Colonization by Burkholderia cepaea or Stenotrophomonas maltophilin
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France